CLINICAL TRIAL: NCT00242749
Title: A Phase 2 Trial to Evaluate ZD1839 (IRESSA) in Combination With Cisplatin & Radiotherapy in Patients With Advanced Head & Neck Carcinoma (Unresectable &Inoperable)
Brief Title: IRESSA in Combination With Cisplatin & Radiotherapy in Patients With Advanced Head & Neck Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0102
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Cancer of Head and Neck
Keywords: Head and Neck Cancer Disease; Head Cancer; Neck Cancer; Cancer of Head; Cancer of Neck; Cancer of the Head; Cancer of the Head and Neck; Cancer of the Neck; Neoplasms, Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Gefitinib; Cisplatin; Radiotherapy

INTERVENTIONS:
Drug: Gefitinib, Cisplatin and Radiotherapy

SUMMARY:
· To evaluate the disease free survival rate at 2 years of patients with advanced head and neck carcinoma treated with ZD1839 250 mg administered once daily in combination with cisplatin and a standard course of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous head and neck carcinoma
2. Extra-laryngeal tumour or laryngeal tumour that is inoperable (not resectable) considered by Head and Neck Cancer Committee
3. Stage III-IV (IVa and IVb) disease
4. Measurable disease according to RECIST criteria
5. Aged 18 years or older
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
7. Normal renal, haematological (neutrophils >1´5 x 109/ L and platelets > 100 x 109/L) and liver function

Exclusion Criteria:

* 1. Previous treatment for initial disease (neck dissection in N3 is allowed) 2. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ 3. Incomplete healing from previous oncologic or other surgery 4. Absolute neutrophil count (ANC) less than 1.5 x 109/ L, or platelets less than 100x 109/L 5. Serum bilirubin greater than 1.25 times the upper limit of reference range (ULRR) 6. In the opinion of the investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease) 7. Serum creatinine greater than 1.25 times the ULRR 8. ALT or AST greater than 2.5 times the ULRR 9. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial 10. Active dermatoses (e.g. psoriasis, eczema) 11. Corneal abnormalities (other than scars, congenital abnormality or corneal tear film), history of dry eye syndrome or ocular surface diseases and neurological disorders 12. Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin or drugs with known corneal toxicity 13. Pregnancy or breastfeeding (women of child-bearing potential) 14. Patient incapacity to reliably follow the treatment or follow up for family, economic or geographical reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47
Dates: Start 2002-12; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Disease-free survival at 2 years

SECONDARY OUTCOMES:
Objective tumour response (CR and PR) at 6 months after the start of treatment based on the Response Evaluation Criteria in Solid Tumours (RECIST) criteria
PFS
Nature, incidence and severity of adverse events (AEs)
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Spain Medical Director, MD, Study Director — AstraZeneca
Locations (4):
- Spain (4):
  - Research Site, Badalona
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Santander